CLINICAL TRIAL: NCT00998439
Title: PEPCAD DES - Treatment of DES-In-Stent Restenosis With SeQuent® Please Paclitaxel Eluting PTCA Catheter
Brief Title: Treatment of Drug-eluting Stent (DES) In-Stent Restenosis With SeQuent® Please Paclitaxel Eluting Percutaneous Transluminal Coronary Angioplasty (PTCA) Catheter
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Klinikum Coburg (Other)
Responsible Party: Harald Rittger, MD, Klinikum Coburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEPCAD DES
Record Dates: First submitted 2009-09-10; First posted 2009-10-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: In-Stent Restenosis
Keywords: in stent restenosis; paclitaxel coated balloon catheter; pepcad; drug eluting balloon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel coated balloon catheter (Experimental)
  Interventions: Device: SeQuent® Please
- uncoated balloon catheter (POBA) (Active Comparator)
  Interventions: Device: SeQuent® II

INTERVENTIONS:
Device: SeQuent® Please — * 6 F, 7 F, or 8 F guiding catheters have to be used
  * after insertion of arterial sheath, apply heparin (7,500-10,000 Units i.a. or i.c. (or 50-100 U/kg body weight))
  * additional dose of 5,000 Units (75 U/kg body weight) if procedure lasts for more than one hour
  * Nitroglycerin (0.2 mg i.c.) prior to first contrast injection
  * ISR must be predilated with uncoated balloon
  * balloon diameter shall be 0.5 mm smaller than the Paclitaxel-eluting balloon intended for use
  * inflation time has to be ≥ 30 sec
  * select balloon with correct stent diameter to achieve a remaining stenosis of ≤ 10 %
  * each Paclitaxel-eluting balloon catheter is allowed for single use only
  * additional inflations and/or aggressive anti-platelet agents for intraluminal defects or haziness
  * if additional balloon is necessary, only uncoated balloon is permitted to avoid overdosing of drug
  Other Names: paclitaxel coated balloon catheter; DEB
  Arms: Paclitaxel coated balloon catheter
Device: SeQuent® II — * 6 F, 7 F, or 8 F guiding catheters have to be used
  * after insertion of arterial sheath, apply heparin (7,500-10,000 Units i.a. or i.c. (or 50-100 U/kg body weight))
  * additional dose of 5,000 Units (75 U/kg body weight) if procedure lasts for more than one hour
  * Nitroglycerin (0.2 mg i.c.) prior to first contrast injection
  * ISR must be predilated with uncoated balloon
  * balloon diameter shall be 0.5 mm smaller than the Paclitaxel-eluting balloon intended for use
  * inflation time has to be ≥ 30 sec
  * select balloon with correct stent diameter to achieve a remaining stenosis of ≤ 10 %
  * each Paclitaxel-eluting balloon catheter is allowed for single use only
  * additional inflations and/or aggressive anti-platelet agents for intraluminal defects or haziness
  * if additional balloon is necessary, only uncoated balloon is permitted to avoid overdosing of drug
  Other Names: uncoated balloon catheter
  Arms: uncoated balloon catheter (POBA)

SUMMARY:
The aim of the study is to assess the efficacy of the Paclitaxel-eluting PTCA - balloon catheter SeQuent® Please to treat in-stent restenoses (ISR) of various drug eluting stents in native coronary arteries with reference diameters between 2.5 mm and ≤ 3.5 mm and lesion lengths ≤ 22 mm. The vessel patency following treatment with SeQuent® Please will be documented in ISR patients that have been treated with the Cypher® or Taxus® drug eluting stent.

DETAILED DESCRIPTION:
Background information

Current treatments for In Stent Restenosis (ISR) are 'uncoated balloon only' angioplasty with conventional balloons (POBA), Bare Metal Stent (BMS) implantations, cutting balloons, rotablation and atherectomy. Their respective results to lower target vessel revascularizations were in part unsatisfactory and often conflicting. Also the temporary use of brachytherapy lead to late lumen loss (LLL) findings in the range from 0.22 ± 0.84 mm. Therefore, brachytherapy to treat ISR has also been abandoned because of the associated delayed endothelialization leading to late thrombosis.

The use of drug eluting stents (DES) to treat ISR lowered restenosis rates in the single digit range. Recently, the use of matrix coated paclitaxel-eluting PTCA balloon catheters (SeQuent® Please, Paccocath Technology®, Bayer/Schering & B.Braun Melsungen AG) was compared to PES in the PEPCAD II trial which showed significantly lower 6-month LLL, 6-month MACE and TVR rates for SeQuent® Please (7.25%) as compared to PES for which the 12-month TVR rate was 19.0% and therefore in agreement with prior studies (ISAR DESIRE). Since these assessments were done in patients with BMS in-stent restenosis, it is of paramount interest to study in-stent restenosis of failed DES implantations since they may cause continued chronic inflammatory responses caused by the non-bioabsorbable polymer in particular once the drug release has ceased.

ELIGIBILITY:
Inclusion Criteria: Patient Related

* Patients with stable angina pectoris (CCS class 1-3) or with unstable angina pectoris (Braunwald class 1-2, A-C) or documented ischemia or with documented silent ischemia
* Patients eligible for coronary revascularization by means of PCI
* Patients suitable for coronary revascularization of any sort (balloon angioplasty, device-assisted balloon-angioplasty, or coronary artery bypass grafting)
* Patients must be ≥ 18 years of age
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 6 months follow-up
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 6 months angiographic follow-up
* Patients must agree to undergo the 1 and 3 year clinical follow-up
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of this trial, e.g., balloon angioplasty by means of the paclitaxel-eluting PTCA-balloon catheter or other suitable devices. The patients, by providing their informed consent, agree to these risks and benefits as stated in the patient informed consent document.

Inclusion Criteria: Lesion Related

* In-stent restenosis or Mehran type III stenoses reaching ≤ 2 mm into the adjacent native vessel of a drug eluting stent (DES), in a native coronary artery (reference vessel between ≥ 2.5 and ≤ 3.5 mm, lesion length ≤ 22 mm as angiographically documented)
* Diameter stenosis pre procedure must be either ≥ 70 % or ≥ 50 % if ischemia corresponding to the target lesion is documented either by exercise stress ECG, stress echocardiography, scintigraphy, MRT, or suspected based on angina pectoris.
* DES in-stent restenosis independent of the the number of metal layers (e.g. restenosed DES following BMS and/or DES implantation(s))

Exclusion Criteria: Patient Related

* Patients with acute (< 24 h) or recent (48 hours) myocardial infarction
* Patients with unstable angina pectoris (Braunwald class 3)
* Patients with severe congestive heart failure
* Patients with severe heart failure NYHA IV
* Patients demonstrating clinical signs of cardiogenic shock at the time of the procedure (systolic blood pressure of less than 80 mmHg requiring inotropic support, IABP and/or fluid challenge)
* Patients with severe valvular heart disease
* Women who are pregnant or lactating patients with life expectancy of less than five years or factors making clinical follow-up difficult
* Patients with another coronary stent previously implanted into the target vessel
* Patients with bleeding diathesis in whom anticoagulation or anti-platelet medication is contraindicated
* Patients who had a cerebral stroke < 6 months prior to the procedure
* Patient participates in other clinical trials involving any investigational device or drug
* Untreated hyperthyroidism
* Patient has presence or history of severe renal failure (GFR < 30ml/min) and is therefore not eligible for angiography. Patient's serum creatinine levels must be documented.
* Post transplantation of any organ or immune suppressive medication
* Other disease to jeopardize follow-up (e.g. malignoma)
* Addiction to any drug or to alcohol
* Patients with any type of surgery during the week preceding the interventional procedure
* Conditions which prevent the intake of the double anti-platelet therapy for three months

Exclusion Criteria: Lesion Related

* Evidence of extensive thrombosis within target vessel before the intervention
* Side branch > 2 mm in diameter originating from the stent
* Bifurcate lesion
* Left main coronary artery stenosis
* Multilesion percutaneous coronary intervention within the same artery (a main artery e.g., LCX and its side branch e.g. OMS are considered as different arteries)
* Percutaneous coronary intervention of venous graft
* Coronary artery occlusions of any type (e.g. acute or chronic)
* In-segment stenosis of the native vessel within the 5 mm adjacent to the stent
* Lesion within 1 mm of vessel origin

Exclusion Criteria: Related to Concomitant Medication

* Patient is intolerant to aspirin and/or the ADP-antagonists clopidogrel or has a history of neutropenia, thrombocytopenia induced by ADP-antagonists, or severe hepatic dysfunction prohibiting the use of clopidogrel
* Patient has leucopoenia (leukocyte count < 109/liter for more than 3 days)
* Patient has neutropenia (ANC < 1000 neutrophils/mm3 for more than 3 days)
* Patient has a history of peptic ulcer or gastric/intestinal bleeding during the past 6 months
* Patient has a history of thrombocytopenia (< 100,000 platelets/mm3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss | 6 months

SECONDARY OUTCOMES:
Occurrence of acute (up to 48 hours), subacute (up to 30 days), and late thrombosis | 3 years
Major adverse cardiac event (MACE) rate | 30 days
Percent in-stent stenosis | 6 months
Percent in-segment stenosis | 6 months
In-stent late loss index | 6 months
Angiographic binary in-stent stenosis rate | 6 months
In-segment late loss index | 6 months
Angiographic binary in-segment stenosis rate | 6 months
Indication for premature follow-up | 6 months
Type of recurrence (Mehran-Classification) | 6 months
Target vessel failure | 6 months
MACE Rate | 6 months
MACE Rate | 1 year
MACE Rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Harald Rittger, MD, Principal Investigator — Klinikum Coburg
Locations (8):
- Germany (8):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Klinikum Bayreuth, Bayreuth
  - Klinikum Coburg, Coburg
  - Klinikum Kulmbach, Kulmbach
  - Herzzentrum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - LMU - Klinikum der Universität München, Munich
  - Klinikum Weiden, Weiden

REFERENCES:
- [Derived] Rittger H, Wohrle J, Brachmann J, Hohenforst-Schmidt W, Schlundt C, Lonke S, von Cranach M, Markovic S, Achenbach S, Waliszewski M. Angiographic patterns of drug-eluting stent restenosis after treatment with drug-coated balloon versus balloon angioplasty: Late lumen loss subgroup analyses of the PEPCAD-DES study. Catheter Cardiovasc Interv. 2016 Oct;88(4):529-534. doi: 10.1002/ccd.26451. Epub 2016 Feb 19. PMID 26893095
- [Derived] Rittger H, Waliszewski M, Brachmann J, Hohenforst-Schmidt W, Ohlow M, Brugger A, Thiele H, Birkemeyer R, Kurowski V, Schlundt C, Zimmermann S, Lonke S, von Cranach M, Markovic S, Daniel WG, Achenbach S, Wohrle J. Long-Term Outcomes After Treatment With a Paclitaxel-Coated Balloon Versus Balloon Angioplasty: Insights From the PEPCAD-DES Study (Treatment of Drug-eluting Stent [DES] In-Stent Restenosis With SeQuent Please Paclitaxel-Coated Percutaneous Transluminal Coronary Angioplasty [PTCA] Catheter). JACC Cardiovasc Interv. 2015 Nov;8(13):1695-700. doi: 10.1016/j.jcin.2015.07.023. PMID 26476609
- [Derived] Rittger H, Brachmann J, Sinha AM, Waliszewski M, Ohlow M, Brugger A, Thiele H, Birkemeyer R, Kurowski V, Breithardt OA, Schmidt M, Zimmermann S, Lonke S, von Cranach M, Nguyen TV, Daniel WG, Wohrle J. A randomized, multicenter, single-blinded trial comparing paclitaxel-coated balloon angioplasty with plain balloon angioplasty in drug-eluting stent restenosis: the PEPCAD-DES study. J Am Coll Cardiol. 2012 Apr 10;59(15):1377-82. doi: 10.1016/j.jacc.2012.01.015. Epub 2012 Feb 29. PMID 22386286